CLINICAL TRIAL: NCT01759888
Title: From Mouse Models to Patients: Development of a Novel 18F-DTBZ PET Imaging as a Biomarker to Monitor Neurodegeneration of PARK6 and PARK8 Parkinsonism
Brief Title: Development of a Novel 18F-DTBZ PET Imaging as a Biomarker to Monitor Neurodegeneration of PARK6 and PARK8 Parkinsonism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, NJI90OKM, Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 100-1926A
Record Dates: First submitted 2013-01-01; First posted 2013-01-03 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-DTBZ for Parkinson's Disease (Experimental): This study will compare the brain uptake of 18F- DTBZ in 60 PD patients, including 20 LRRK2 G2385R, 20 PARK6, and 20 idiopathic PD. Subjects will be evaluated sequentially with 18F-DTBZ during a 36 month period. 18F-DTBZ PET scans will be performed twice, at baseline, and 24 (21~27) months following the start of their participation in the study.
  Interventions: Drug: 18F-DTBZ

INTERVENTIONS:
Drug: 18F-DTBZ — Subjects will receive a single i.v. administration of approximately 10 mCi 18F-FP-(+)-DTBZ (10 nmole FP-(+)-DTBZ) immediately prior to each scan.
  The proposed dose for this study is based on our phase I study. At the proposed human dose of 10 mCi, the whole body effective dose (ED) will be approximately 680 mrem. The estimated human ED is expected to be comparable to or below the range of other approved brain imaging agents, such as 18F-FDG.

SUMMARY:
The primary objective of this protocol is to access the utility of 18F-DTBZ PET imaging as an in vivo biomarker to monitor neurodegeneration of both PD mouse models and PD patients. Secondary, the investigators will analyze progression rate of genetic-proving PARK8 and PARK6 patients who have homogeneous phenotype and genotype by 18F-DTBZ PET imaging.

DETAILED DESCRIPTION:
Total of 60 patients, 20 LRRK2 G2385R, 20 PARK6, and 20 idiopathic PD, will be recruited. Subjects will be evaluated sequentially with 18F-DTBZ during a 36 month period. 18F-DTBZ PET scans will be performed twice, at baseline, and 24 (21~27) months following the start of their participation in the study. Subjects will receive a single i.v. administration of approximately 10 mCi 18F-DTBZ immediately prior to imaging. Whitney test will be used to compare the mean standard uptake value ratio (SUVR) values between groups. The decline rate of VMAT2 density will be calculated by comparing the SUVRs of age-matched healthy subjects from our previous studies. Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, each subject will have 3 visits in each scan (total 6 visits in this study), as one screening visit, one imaging visit, and one safety evaluation visit.

Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders and 20~80 years old.
2. Written and dated informed consent by self or by legal representative, to be obtained before any of the study procedures.
3. Twenty PD patients were proved carrying LRRK2 G2385R mutation by our genetic laboratory. Patients didn't have other mutations that may contribute to the parkinsonism, such as LRRK2 G2019S, LRRK2 R1628P, PARK2, PARK6, and SCA2.
4. Twenty PARK6 PD patients were proved carrying PINK1 mutation by our genetic laboratory. Patients didn't have other mutations that may contribute to the parkinsonism, such as LRRK2, PARK2, and SCA2.
5. Twenty idiopathic PD patients were proved that they did not carry any known mutations, which may contribute to the parkinsonism, such as LRRK2, PARK2, PARK6, and SCA2. The age of disease onset should be more than 50 years, and no known familial history of parkinsonism or spinocerebellar atrophy.
6. All the subjects should be fulfilled the UK Parkinson's Disease Society Brain Bank criteria of "possible" or "probable" PD.

Exclusion Criteria:

1. Pregnant or becoming pregnant during the study or current breast feeding.
2. Any subject who has a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.

   1. Clinically significant hepatic, renal, pulmonary, metabolic, or endocrine disturbances, especially thyroid disease.
   2. Current clinically significant cardiovascular disease. (cardiac surgery or myocardial infarction within the last 6 months; unstable angina; decompensated congestive heart failure; significant cardiac arrhythmia; congenital heart disease.
3. History of drug or alcohol abuse within the last year, or prior prolonged hi story of abuse.
4. History or presence of QTc prolongation.
5. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
6. Any documented abnormality in the brain by CT or MRI of brain, which might contribute to the motor function, such as hydrocephalus, multiple infarction and encephalomalacia, will be excluded. Mild cortical atrophy and non-specific white matter changes will be allowed.
7. Any evidence of secondary parkinsonism (multiple infarcts, intoxication, and hydrocephalus, etc).
8. General PET exclusion criteria.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To calculate the decline rate of striatal 18F-FP-(+)-DTBZ binding and to evaluate whether the degenerative rate differs between idiopathic PD patients and genetic-proving PARK6/PARK8 patients | 2 years
  The annual decline rate of striatal 18F-DTBZ SUVRs (specific uptake value ratios) in PD patients carrying LRRK2 G2385R mutation, PARK6 patients, and patients with idiopathic PD, respectively.

SECONDARY OUTCOMES:
To analyze the correlation between decline rate of 18F-FP-(+)-DTBZ uptake and clinical severity, and access the feasibility of 18F-DTBZ PET imaging as an in vivo biomarker to monitor neurodegeneration in PD | 1 year
  To analyze the correlation between 18F-FP-(+)-DTBZ annual decline rate and the progression rate of clinical motor scores/non-motor scores/ neuropsychiatric tests in each group. Furthermore, to access the utility of 18F-DTBZ PET imaging as an in vivo biomarker to monitor neurodegeneration in PD patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memory Hpspital, Taoyuan District, Taiwan